CLINICAL TRIAL: NCT06244238
Title: A Study on the Relationship Between Job Satisfaction and Retention Intentions of Emergency Room Nurses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202311079RINB
Record Dates: First submitted 2024-01-11; First posted 2024-02-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: A Study on the Relationship Between Job Satisfaction and Retention Intentions of Emergency Room Nurses
Keywords: Emergency Room Nurses 、 Job Satisfaction 、Retention Intentions
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency Nurse: 1. Employed in an urgent care unit.
  2. Holds a nursing or registered nurse license.
  3. Currently engaged in nursing duties.
  4. Has a minimum of three months of nursing service in this hospital.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
Based on a survey conducted by the Nursing and Health Care Bureau of the Ministry of Health and Welfare in 2023, which investigated the recruitment and turnover rates of nursing personnel in 479 hospitals of different levels, the results revealed that the recruitment of nursing personnel was exceedingly challenging. The difficulty levels varied, with medical centers at 80%, regional hospitals at 67.9%, and district hospitals at 43.37%. Additionally, the turnover rates of nursing personnel were notably high, with medical centers at 10.21%, regional hospitals at 11.17%, and district hospitals at 14.52%. These rates all exceeded 10%, which means that, on average, one out of every ten nursing personnel resigned (Nursing and Health Care Bureau, Ministry of Health and Welfare, 2023).

This study aims to investigate the relationship between job satisfaction and retention intention among emergency room nursing personnel in a regional teaching hospital in Yunlin County. In the fiscal year 2023, the unit experienced an alarming turnover rate of approximately 82% among newly hired personnel. Therefore, the study intends to conduct further research and exploration into the job satisfaction and retention intention of emergency room nursing personnel.

The primary objectives of the research include examining the correlation between the demographic characteristics of emergency room nurses and their job satisfaction, the correlation between the demographic characteristics of emergency room nurses and their retention intention, and the correlation between job satisfaction and retention intention among emergency room nurses.

The study's subjects are nurses or nursing staff employed in the emergency department. The research is conducted through the distribution of questionnaires, and all responses are collected anonymously. The questionnaire is structured into three main sections: the first section covers demographic characteristics, the second section addresses job satisfaction items, and the third section focuses on retention intention items.

Upon collecting and encoding the data, the information will be compiled, and statistical analysis will be performed using Excel and SPSS version 25.0 statistical software to validate various research hypotheses.

The expected outcome of the study is a positive relationship between job satisfaction and retention intention among emergency room nurses, indicating that job satisfaction influences retention intention.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Nurse
* Employed in an urgent care unit.
* Holds a nursing or registered nurse license.
* Currently engaged in nursing duties.
* Has a minimum of three months of nursing service in this hospital.

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Nurse meeting the aforementioned qualification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-03 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
The questionnaire | 2024/01/15-2024/02/29
  The research questionnaire is structured into four main sections: The first section covers demographic information; the second section addresses job satisfaction; and the third section explores intentions related to nursing retention. In the first part, demographic information is gathered from respondents, including gender, age, education level, marital status, number of children, years of work experience, job position, advanced qualifications, and work shift. The second part focuses on job satisfaction with a total of 31 questions, while the third part delves into nursing retention intentions with a set of 5 questions.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Tianwan, Tianwan, Taiwan
  - Tiawan, Tianwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data collected for this study is intended solely for the purpose of this research.

REFERENCES:
- See also: National Union of Taiwan Nurses' Associations - Nursing Personnel Statistics for the Taiwan and Fujian Regions, August 2023. — https://www.nurse.org.tw/publicUI/H/H10201.aspx?arg=8DBAD2670041C77005